CLINICAL TRIAL: NCT07318636
Title: An Open-Label, Single-Arm Study Evaluating the Safety and Efficacy of NK010 Cell Injection Combined With PD-1 Antibody and Platinum-Based Chemotherapy as Neoadjuvant Therapy in Patients With Resectable Non-Small Cell Lung Cancer
Brief Title: NK-cell Therapy Combined With PD-1 Antibody and Platinum-Based Chemotherapy as Neoadjuvant Therapy in Resectable NSCLC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Shanghai NK Cell Technology Co., LTD (Industry)
Responsible Party: Principal Investigator, Jianxing He, President, Guangzhou Institute of Respiratory Health, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK010-IIT-NSCLC-01
Record Dates: First submitted 2025-12-16; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Resectable Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NK010 + PD-1 Antibody + Platinum-Based Chemotherapy (Experimental): Participants will receive neoadjuvant therapy for a total of 3 cycles, with each cycle lasting 3 weeks. NK010 cell injection will be administered in combination with a PD-1 antibody and platinum-based chemotherapy. After completing 3 cycles of treatment, participants will undergo surgical resection, followed by pathological assessment to evaluate outcomes such as major pathological response (MPR), pathological complete response (pCR), and R0 resection rate. NK010 administration will be evaluated at three planned dose levels.
  Interventions: Drug: PD-1 antibody; Biological: NK010

INTERVENTIONS:
Drug: PD-1 antibody — The PD-1 antibody will be administered intravenously in combination with NK010 cell injection and platinum-based chemotherapy during the neoadjuvant treatment phase.
Biological: NK010 — NK010 is an allogeneic, off-the-shelf natural killer (NK) cell product derived from peripheral blood. NK010 will be administered intravenously in combination with a PD-1 antibody and platinum-based chemotherapy during the neoadjuvant treatment phase.

SUMMARY:
This open-label, single-arm study is designed to evaluate the safety and preliminary efficacy of NK010 cell injection combined with a PD-1 antibody and platinum-based chemotherapy as neoadjuvant therapy in patients with resectable non-small cell lung cancer (NSCLC). The study aims to assess the safety profile, feasibility of administration, and potential antitumor activity of this combination regimen.

DETAILED DESCRIPTION:
Participants with histologically or cytologically confirmed, resectable non-small cell lung cancer (NSCLC) will receive a neoadjuvant regimen consisting of NK010 cell injection, an anti-PD-1 antibody, and standard platinum-based doublet chemotherapy.

The primary objective of this study is to assess the safety and feasibility of this combination regimen in the preoperative setting. Secondary objectives include the exploration of potential antitumor activity. The study utilizes a sequential dose-escalation design, with NK010 administered at three planned dose levels.

Following neoadjuvant therapy and surgical resection, postoperative adjuvant therapy will be administered at the investigator's discretion in accordance with standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and voluntarily sign the written informed consent form (ICF).
* Male or female patients aged ≥18 years.
* Histologically and/or cytologically confirmed resectable stage IB to IIIA non-small cell lung cancer (NSCLC) according to AJCC 8th edition.
* Treatment-naïve NSCLC (no prior systemic anticancer therapy).
* No sensitizing EGFR mutations (exon 19 deletion, exon 21 L858R) and no ALK gene rearrangement.
* At least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Estimated life expectancy of more than 6 months.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Adequate bone marrow, liver, and renal function.
* Female participants of childbearing potential must have a negative pregnancy test prior to initiation of study treatment.

Exclusion Criteria:

* Prior receipt of any systemic anticancer therapy.
* Known sensitizing EGFR mutations or ALK gene rearrangements.
* Active, known, or suspected autoimmune disease.
* Interstitial lung disease.
* Any medical condition, therapy, or laboratory abnormality that, in the opinion of the investigator, could confound the study results, interfere with the participant's ability to comply with study procedures, or is not in the best interest of the participant.
* Locally advanced unresectable or metastatic NSCLC.
* Major cardiovascular events, unstable arrhythmia, or unstable angina within 3 months prior to study treatment initiation.
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use effective contraception during the study.
* Any other condition judged by the investigator to make the participant unsuitable for clinical trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 1 year after first dose of NK010
  Number of subjects experiencing adverse events, and the frequency and severity of adverse events. The type, frequency, onset, and severity of treatment-emergent adverse events (TEAEs) will be assessed in accordance with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Dose Limiting Toxicities (DLTs) | Up to 21 days after first dose of NK010
  Identification of DLTs to determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Major pathological response (MPR) | Within 6 weeks after completion of neoadjuvant therapy
  The MPR rate will be reported as the proportion of participants achieving MPR among all participants who undergo surgical resection.
Pathological complete response (pCR) | Within 6 weeks after completion of neoadjuvant therapy
  The pCR rate will be reported as the proportion of participants achieving pCR among all participants who undergo surgical resection.
R0 Resection Rate | Within 6 weeks after completion of neoadjuvant therapy
  The proportion of participants who achieve complete surgical tumor resection
Objective Response Rate (ORR) | Up to preoperative assessment (approximately 12 weeks from treatment initiation)
  ORR is defined as the proportion of participants achieving a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria, as assessed by radiologic imaging after completion of neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No